CLINICAL TRIAL: NCT02513147
Title: HIV Reservoir Dynamics After Switching to Dolutegravir in Patients With Two NRTI and a Protease Inhibitor Based Regimen. A Phase IV Open Randomized Trial
Brief Title: HIV Reservoir Dynamics After Switching to Dolutegravir in Patients on a PI and 2 NRTI Based Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: University Hospital, Ghent (Other); IrsiCaixa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDOOR
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: HIV-1
MeSH Terms: interventions — dolutegravir; fosamprenavir; Atazanavir Sulfate; Lopinavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 NRTI+ Dolutegravir (Experimental): 22 patients will be treated with 2 NRTI+Dolutegravir 50 mg during 24 weeks
  Interventions: Drug: Dolutegravir; Drug: 2 NRTI
- 2 NRTI + PI (Active Comparator): 22 patients will be treated with 2 NRTI + PI during 24 weeks
  Interventions: Drug: PI; Drug: 2 NRTI

INTERVENTIONS:
Drug: Dolutegravir
  Arms: 2 NRTI+ Dolutegravir
Drug: PI — (Fosamprenavir, atazanavir, lopinavir or darunavir) boosted with 100 mg of ritonavir, or atazanavir (400 mg / d) not boosted with ritonavir,if the 2 NRTIs are abacavir + Lamivudine
  Other Names: Fosamprenavir, atazanavir, lopinavir or darunavir
  Arms: 2 NRTI + PI
Drug: 2 NRTI
  Arms: 2 NRTI+ Dolutegravir
Drug: 2 NRTI
  Other Names: 2NRTI
  Arms: 2 NRTI + PI

SUMMARY:
The purpose of this study is to assess changes in viral reservoir after changing IP/r to dolutegravir in HIV-1 infected patients maintaining undetectable viral load on Antiretroviral Therapy (ART).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients infected with HIV-1
* HIV RNA <50 copies / mL for ≥ 1 year with stable ART regimen (≥ 3 months) based on 2 NRTI and PI (Fosamprenavir, atazanavir, lopinavir or darunavir) boosted with 100 mg of ritonavir, or atazanavir (400 mg / d) not boosted with ritonavir, if the 2 NRTIs are abacavir + Lamivudine
* CD4 + lymphocytes > 200 / mm3
* Signature of voluntary informed consent
* A woman may be eligible to enter and participate in the study if:

  1. No reproductive potential-defined as post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of getting pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.
  2. It is in childbearing age with a negative pregnancy test on the day of screening and on Day 1 and agrees to use one of the following contraceptive methods to prevent pregnancy:

     * Complete abstinence from penis-vaginal from 2 weeks prior to administration of investigational product, throughout the study, and for at least 2 weeks after discontinuation of all study drugs;
     * Double barrier method (male / spermicidal condom, male condom / diaphragm, diaphragm / spermicide);
     * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion)
     * Male sterilization confirmed before the entry of the female subject in the study, and that this man is the only sexual partner for women
     * Approved hormonal contraception
     * Any other method with published data show that the expected failure rate is <1% per year.

Exclusion Criteria:

* Prior virologic failure with an integrase inhibitor
* Acquired Immune Deficiency Syndrome (AIDS)-defining illness in the last 48 weeks
* Glomerular filtration rate <50 mL / min, estimated by Chronic Kidney Disease Epidemiology (CKD-EPI) formula
* Alanine aminotransferase (ALT) ≥5 times the Upper Limit Normal (ULN) or ALT ≥3 X ULN and total bilirubin ≥1,5 ULN (with> 35% direct bilirubin) and / or unstable liver disease (with the presence of ascites, hepatic encephalopathy, hypoalbuminemia, esophageal varices or persistent jaundice) or known biliary disorders excluded Gilbert syndrome or asymptomatic lithiasis) .
* Positive for hepatitis B (HBsAg +) or need for Hepatitis C Virus (HCV) treatment during the study .
* Subjects with severe hepatic impairment (Child Pugh Class C).
* Patients unable to understand the study protocol or any other condition that in the investigator's opinion could jeopardize compliance with the protocol
* Pregnant or breast-feeding
* History or presence of allergy to any of the study drugs or their components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in mean of Long Terminal repeat (2LTR) in lymphocytes T Cluster of Differentiation 4+ (CD4 +) in peripheral blood obtained at week 1 of the study compared to day 0 | 1 week
Changes in mean of Long Terminal repeat (2LTR) in lymphocytes T Cluster of Differentiation 4+ (CD4 +) in peripheral blood obtained at week 2 of the study compared to day 0 | 2 weeks
Changes in mean of Long Terminal repeat (2LTR) in lymphocytes T Cluster of Differentiation 4+ (CD4 +) in peripheral blood obtained at week 4 of the study compared to day 0 | 4 weeks
Changes in mean of Long Terminal repeat (2LTR) in lymphocytes T Cluster of Differentiation 4+ (CD4 +) in peripheral blood obtained at week 12 of the study compared to day 0 | 12 weeks
Changes in mean of Long Terminal repeat (2LTR) in lymphocytes T Cluster of Differentiation 4+ (CD4 +) in peripheral blood obtained at week 24 of the study compared to day 0 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain